CLINICAL TRIAL: NCT02488044
Title: A Phase 1/2 Open-label Study in Patients With Arginase I Deficiency to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous AEB1102
Brief Title: A Phase 1/2 Study of AEB1102 in Patients With Arginase I Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeglea Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAEB1102-101A
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Arginase I Deficiency; Hyperargininemia
MeSH Terms: conditions — Hyperargininemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AEB1102 (Experimental): AEB1102, modified human Arginase I administered IV Part 1 Each patient may receive up to 7 doses given up to every other week over a maximum of 14 weeks.
  Part 2 Each patient will receive up to 8 weeks of repeat-dose therapy.
  Interventions: Drug: AEB1102

INTERVENTIONS:
Drug: AEB1102 — modified human arginase I
  Other Names: Co-ArgI-PEG

SUMMARY:
A Phase 1/2 Open-label Study in Patients with Arginase I Deficiency to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous AEB1102. This study is designed to evaluate the safety and tolerability of IV administration of AEB1102 for the treatment of pediatric and adult patients with Arginase I deficiency and hyperargininemia. This study will be conducted in 2 parts: Part 1 (Single Ascending Dose Escalation) and Part 2 (Repeated Dosing). Each part will be preceded by a baseline assessment of arginine levels. All patients who participate in Part 1 may continue AEB1102 dosing in Part 2 if they qualify for continued dosing. A data safety monitoring board (DSMB) will provide independent review of study safety data and recommend whether the sponsor should continue the study as planned, modify the study protocol, or discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Arginase I deficiency
* Adequate organ function: Hgb ≥ 10 g/dL, ANC ≥ 1.5 x 109/L, plt count ≥ 100,000/µL; liver transaminase levels ≤ 2.5x ULN, total bilirubin ≤ 2.0 mg/dL; serum creatinine <1.5 x ULN
* If female and of child-bearing potential, has a negative serum pregnancy test within 7 days before enrollment
* If a sexually active (male or female), must be surgically sterile, post-menopausal (female), or must agree to use a physician-approved method of birth control during the study and for a minimum of 30 days after the last study drug administration
* Patient or legal guardian is able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures and continuation of prescribed diet without modification) prior to any screening procedures

Exclusion Criteria:

* Transfusion of ≥ 2 u RBC within 60 days
* Active infection requiring systemic treatment
* Known infection with HIV, Hep B or Hep C
* Severe hyperammonemia requiring hospitalization within 14 days. Had more than one episode of hyperammonemia requiring hospitalization within the 30 days prior to enrollment.
* Current uncontrolled hyperammonemia
* Has a history of hypersensitivity to PEG or any other component of the AEB1102 (Co-ArgI-PEG) formulation
* If female, is lactating or breast feeding

PART 2 INCLUSION CRITERION:

1. Did not experience any safety or tolerability event in Part 1 which would preclude continued participation and dosing of AEB1102

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | weekly throughout the study, up to 14 weeks
  Includes significant changes in hematology, chemistry and coagulation laboratory studies as well as in physical exam and vital signs

SECONDARY OUTCOMES:
Number of subjects with a decrease from baseline in plasma arginine level | Baseline to 2, 4, 6, 8 weeks
Pharmacokinetic profile including Cmax, AUC, Tmax, T1/2 for each subject | At 15 min, 1, 2, 4, 8, 12, 24, 48, 72, and 120 hours following dose escalation
Number of subjects with a decrease from baseline in plasma guanidino compound levels | Baseline to 2, 4, 6, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Josie Gayton, Study Director — Aeglea Biotherapeutics, Inc.
Locations (9):
- United States (6):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida, Gainesville, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UTSW, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Centro Hospitalar S. Joao, Porto, Portugal
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Background] Crombez EA, Cederbaum SD. Hyperargininemia due to liver arginase deficiency. Mol Genet Metab. 2005 Mar;84(3):243-51. doi: 10.1016/j.ymgme.2004.11.004. Epub 2004 Dec 19. PMID 15694174
- [Background] Glazer ES, Stone EM, Zhu C, Massey KL, Hamir AN, Curley SA. Bioengineered human arginase I with enhanced activity and stability controls hepatocellular and pancreatic carcinoma xenografts. Transl Oncol. 2011 Jun;4(3):138-46. doi: 10.1593/tlo.10265. Epub 2011 Jun 1. PMID 21633669
- [Derived] Diaz GA, Schulze A, McNutt MC, Leao-Teles E, Merritt JL 2nd, Enns GM, Batzios S, Bannick A, Zori RT, Sloan LS, Potts SL, Bubb G, Quinn AG. Clinical effect and safety profile of pegzilarginase in patients with arginase 1 deficiency. J Inherit Metab Dis. 2021 Jul;44(4):847-856. doi: 10.1002/jimd.12343. Epub 2021 Jan 26. PMID 33325055